CLINICAL TRIAL: NCT05345405
Title: Improving Social Support Quality Among Survivors Seeking Acute Post-Rape Care: Testing a Supporter-Targeted Intervention
Brief Title: Clinical Trial of a Supporter-Targeted Intervention to Improve Outcomes in Recent Sexual Assault Survivors
Acronym: CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Emily Dworkin, Assistant Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00011982
Record Dates: First submitted 2022-04-06; First posted 2022-04-25 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Stress Disorders, Post-Traumatic; Helping Behavior; Help-Seeking Behavior; Stress; Relationship, Social; Sexual Assault; Sexual Violence; Social Interaction
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Helping Behavior; Help-Seeking Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dyadic CARE (Active Comparator): Participants will receive dyadic CARE following baseline and will complete self-report assessments at post-session-1, Month 1, Month 2, and Month 3.
  Interventions: Behavioral: Dyadic CARE
- Supporter-Only CARE (Active Comparator): Participants will receive supporter-only CARE following baseline and will complete self-report assessments at post-session-1, Month 1, Month 2, and Month 3.
  Interventions: Behavioral: Supporter-Only CARE
- Waitlist Control (No Intervention): After completing baseline, participants will be invited to schedule a CARE session in 3 months (i.e., after the completion of all study assessments). The version of CARE received at that point will be selected by the survivor. Participants will complete self-report assessments at post-session-1, Month 1, Month 2, and Month 3.

INTERVENTIONS:
Behavioral: Dyadic CARE — Dyadic CARE involves two telehealth sessions with a clinician, the survivor, and a supporter of the survivor's choice. Session content uses cognitive-behavioral strategies (e.g., encouraging non-avoidance) to encourage communication and improve supporters' responses in trauma-related conversations. Between sessions, both the survivor and the supporter are instructed to review session content and have guided discussions with the assistance of a workbook.
  Arms: Dyadic CARE
Behavioral: Supporter-Only CARE — Supporter-only CARE involves two telehealth sessions with a clinician and a supporter of the survivor's choice, without the survivor present. Session content uses cognitive-behavioral strategies (e.g., encouraging non-avoidance) to encourage communication and improve supporters' responses in trauma-related conversations. Between sessions, both the survivor and the supporter are instructed to review session content and have guided discussions with the assistance of a workbook.
  Arms: Supporter-Only CARE

SUMMARY:
Communication and Recovery Enhancement (CARE) is a 2-session early intervention for survivors of recent sexual assault and their supporters that aims to improve supporters' ability to respond effectively. The goal of this pilot trial is to understand the acceptability and preliminary efficacy of two versions of CARE: a version in which survivors and supporters attend both sessions together (dyadic CARE) and a version in which supporters attend sessions alone (supporter-only CARE). Survivors aged 14+ with elevated posttraumatic stress symptoms will enroll with a supporter of their choosing. Dyads will be randomized to dyadic CARE, supporter-only CARE, or waitlist control, and will complete self-report assessments at baseline, post-session-1, and follow-ups (1, 2, and 3 months post-baseline). Results will be used to inform future changes to CARE and determine whether a fully-powered randomized controlled trial is warranted.

ELIGIBILITY:
Inclusion Criteria (Survivors):

* Age 14+ years
* Can speak/read English or Spanish
* Have access to a Zoom-capable device
* Screened for eligibility within 10 weeks of sexual assault, defined as any unwanted, distressing sexual contact (e.g., unwanted touching, coerced sexual activity, rape)
* Able to attend first study session within 2 weeks of screening
* Elevated PTSD symptoms at screening as operationalized by a Primary Care PTSD Screen score of 2/5 or above
* Able to identify an eligible supporter
* Have a way to receive survey links and complete surveys privately (i.e., without potential device or account access by the supporter)

Inclusion Criteria (Supporters):

* Age 14+ years
* Can speak/read English or Spanish
* Have access to a Zoom-capable device
* Able to attend first study session within 2 weeks of survivor's screening
* Are in contact with the survivor at least once a week
* In the opinion of the survivor, are able to make an independent decision about whether or not to participate in the study
* Have a way to receive survey links and complete surveys privately (i.e., without potential device or account access by the survivor)

Exclusion Criteria (Survivors):

* Active psychosis
* Active suicidal intent

Exclusion Criteria (Supporters):

* Perpetrated the sexual assault
* Engaged in severe past-year violence or abuse (as defined by the survivor) against the survivor
* The survivor has not told the supporter about the sexual assault at the time of screening and was not already planning to tell the supporter
* In the opinion of the survivor, relational conflict exists between the survivor and supporter that potentially could be exacerbated by program participation

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily R Dworkin, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington School of Medicine, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be archived in the National Archive of Criminal Justice Data. No direct or indirect identifiers will ever be included in the archived dataset. We will submit study instruments and data collection forms, project reports describing our methods, and Institutional Review Board documentation (including copies of consent forms). A syntax file will include (1) recoding of reverse-scored items; (2) calculation of scale scores; (3) addition of a filter variable indicating any cases not included in any final analyses and the corresponding reason for exclusion; and (5) variable and value labels. Technical documentation for the dataset will include variable codebooks with full study instruments and citations, naming conventions, missing value designations, value labels, known data anomalies, and a data user guide.
Supporting Information: Study Protocol, ICF, Analytic Code

REFERENCES:
- [Derived] Dworkin ER, Ruzek JI, Cordova MJ, Fitzpatrick S, Merchant L, Stewart T, Santos JP, Mohr J, Bedard-Gilligan M. Supporter-focused early intervention for recent sexual assault survivors: Study protocol for a pilot randomized clinical trial. Contemp Clin Trials. 2022 Aug;119:106848. doi: 10.1016/j.cct.2022.106848. Epub 2022 Jul 9. PMID 35817294

RESULTS

PARTICIPANT FLOW:
Groups:
- Dyadic CARE: Dyads randomized to receive dyadic CARE. Dyadic CARE involved both dyad members attending 2 sessions and completing a workbook together. Session 1 typically occurred immediately following baseline/randomization (maximum: 2 weeks later). Session 2 typically occurred 2 weeks after Session 1 (maximum: 4 weeks later).
- Supporter-Only CARE: Dyads randomized to receive supporter-only CARE. Supporter-only CARE involved the supporter attending 2 sessions and completing a workbook with the survivor. Session 1 typically occurred immediately following baseline/randomization (maximum: 2 weeks later). Session 2 typically occurred 2 weeks after Session 1 (maximum: 4 weeks later).
- Waitlist Control: Dyads randomized to receive waitlist CARE (invited to complete the CARE version of the survivor's choice following the completion of study measures)
Period: Overall Study
Arm/Group | Dyadic CARE | Supporter-Only CARE | Waitlist Control
Started | 42 (21 survivors and 21 supporters started) | 44 (22 survivors and 22 supporters started) | 42 (21 survivors and 21 supporters started)
Completed | 40 (20 survivors and 20 supporters completed) | 42 (21 survivors and 21 supporters completed) | 41 (21 survivors and 20 supporters completed)
Not Completed | 2 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Did not meet eligibility criteria | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dyadic CARE (Survivors): Survivors randomized to receive dyadic CARE (both dyad members attended both sessions and completed a workbook together)
- Supporter-Only CARE (Survivors): Survivors randomized to receive supporter-only CARE (only the supporter attended both sessions; the dyad completed a workbook together)
- Waitlist Control (Survivors): Survivors randomized to receive waitlist CARE (invited to complete the CARE version of their choice following the completion of study measures)
- Dyadic CARE (Supporters): Supporters randomized to receive dyadic CARE (both dyad members attended both sessions and completed a workbook together)
- Supporter-Only CARE (Supporters): Supporters randomized to receive supporter-only CARE (only the supporter attended both sessions; the dyad completed a workbook together)
- Waitlist Control (Supporters): Supporters randomized to receive waitlist CARE (invited to complete the CARE version of the survivor's choice following the completion of study measures)
- Total: Total of all reporting groups
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors) | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters) | Total
Number analyzed (Participants) | 21 | 22 | 21 | 21 | 22 | 21 | 128
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: One participant did not report their age. Two participants were withdrawn by researchers for not meeting eligibility and were not included in analyses.
  Years
    number analyzed (Participants) | 21 | 21 | 21 | 21 | 21 | 20 | 125
    (all) | 26.48 (9.56) | 23.24 (6.07) | 25.52 (9.32) | 32.48 (10.75) | 37.52 (15.38) | 30.80 (11.87) | 29.33 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant did not report sex. Two participants were withdrawn by researchers for not meeting eligibility and were not included in analyses.
  Participants
    number analyzed (Participants) | 20 | 21 | 21 | 21 | 21 | 21 | 125
    Female | 19 | 18 | 20 | 13 | 16 | 16 | 102
    Male | 1 | 3 | 1 | 8 | 5 | 5 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two participants were withdrawn by researchers for not meeting eligibility and were not included in analyses.
  Participants
    number analyzed (Participants) | 21 | 21 | 21 | 21 | 21 | 21 | 126
    Hispanic or Latino | 4 | 5 | 4 | 17 | 18 | 18 | 66
    Not Hispanic or Latino | 17 | 16 | 17 | 4 | 3 | 3 | 60
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two participants were withdrawn by researchers for not meeting eligibility and were not included in analyses.
  Participants
    number analyzed (Participants) | 21 | 21 | 21 | 21 | 21 | 21 | 126
    American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Asian | 5 | 6 | 4 | 5 | 6 | 4 | 30
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 1 | 0 | 0 | 2 | 0 | 1 | 4
    White | 7 | 8 | 12 | 9 | 10 | 13 | 59
    More than one race | 5 | 3 | 3 | 2 | 1 | 0 | 14
    Unknown or Not Reported | 3 | 3 | 2 | 3 | 4 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Survivor Satisfaction With Intervention at 1 Month Post-baseline (Self Report)
Description: Sum score on Client Satisfaction Scale, completed by survivor. Range: 8 to 32; higher scores indicate greater satisfaction
Time Frame: 1 month
Population: 2 participants did not complete this scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors)
Number analyzed (Participants) | 19 | 21
score on a scale | 28.37 (3.39) | 27.71 (3.51)

2. Primary Outcome: Supporter Satisfaction With Intervention at 1 Month Post-baseline (Self Report)
Description: Sum score on Client Satisfaction Scale, completed by supporter. Range: 8 to 32; higher scores indicate greater satisfaction
Time Frame: 1 month
Population: 2 participants did not complete this scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters)
Number analyzed (Participants) | 20 | 20
score on a scale | 29.79 (2.65) | 29.60 (2.28)

3. Primary Outcome: Change in Survivor Knowledge at 1 Month Post-baseline (Self Report)
Description: Sum score on a knowledge questionnaire reflecting CARE concepts, completed by the survivor. Range: 8 to 40; higher scores indicate more knowledge about CARE concepts.
Time Frame: Baseline, 1 month
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 17 | 20 | 20
score on a scale | 3.24 (3.70) | 0.20 (3.47) | 0.61 (4.75)

4. Primary Outcome: Change in Supporter Knowledge at 1 Month Post-baseline (Self Report)
Description: Sum score on a knowledge questionnaire reflecting CARE concepts, completed by the supporter. Range: 9 to 45; higher scores indicate more knowledge about CARE concepts.
Time Frame: Baseline, 1 month
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 18 | 19 | 18
Points | 4.61 (2.93) | 4.84 (3.55) | 0.33 (2.54)

5. Primary Outcome: Change in Survivor Confusion About Help-seeking Behavior at 1 Month Post-baseline (Self Report)
Description: Sum score on 4-item measure created for this study, completed by survivor. Range: 4 to 20; higher scores indicate greater confusion.
Time Frame: Baseline, 1 month
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 21 | 21
score on a scale | -2.21 (4.04) | -1.14 (3.64) | 0.86 (4.50)

6. Primary Outcome: Change in Supporter Confusion About Helping Behavior at 1 Month Post-baseline (Self Report)
Description: Sum score on the Confusion subscale of the Impact on Friends scale, completed by supporter. Range: 6 to 30; higher scores indicate greater confusion about helping behavior.
Time Frame: Baseline, 1 month
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | -4.35 (3.88) | -3.70 (3.42) | -1.85 (3.23)

7. Primary Outcome: Survivor Disclosure Frequency to Supporter at 1 Month Post-baseline (Self Report)
Description: Single item representing frequency of disclosures to supporter in past month, completed by survivor, adapted from the Early Intervention Clinic Disclosure scale. Survivor will input a numerical response representing number of disclosures. Higher scores indicate more frequent disclosure.
Time Frame: 1 month
Population: Participants were excluded if they did not complete this scale.
Measure: Mean (Standard Error); unit: number of disclosures
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 21 | 21 | 21
number of disclosures | 2.67 (0.21) | 3.02 (0.21) | 2.66 (0.21)

8. Primary Outcome: Supporter Overt Hostile Reactions to Disclosure at 1 Month Post-baseline (Informant Report)
Description: Sum score on Turning Against subscale of the Social Reactions Questionnaire - Shortened, completed by survivor in reference to supporter's reactions in past month. Range: 0 to 24; higher scores indicate more frequent hostile negative reactions.
Time Frame: 1 month
Population: Only assessed among survivors reporting past-month disclosure to the supporter
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 15 | 18 | 17
score on a scale | 1.41 (0.53) | 2.96 (0.49) | 2.49 (0.50)

9. Primary Outcome: Supporter Subtly Unsupportive Reactions to Disclosure at 1 Month Post-baseline (Informant Report)
Description: Sum score on Unsupportive Acknowledgment subscale of the Social Reactions Questionnaire - Shortened, completed by survivor in reference to supporter's reactions in past month. Range: 0 to 24; higher scores indicate more frequent subtly unsupportive reactions.
Time Frame: 1 month
Population: Only assessed among survivors reporting past-month disclosure to the supporter
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 15 | 18 | 17
score on a scale | 2.04 (0.57) | 2.23 (0.52) | 3.34 (0.54)

10. Primary Outcome: Change in Supporter Responsiveness at 1 Month Post-baseline (Informant Report)
Description: Sum score on the Responsiveness subscale of the Perceived Responsiveness and Insensitivity scale, completed by survivor in reference to past month. Range: 0 to 40; higher scores indicate greater responsiveness.
Time Frame: Baseline & 1 month
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 21 | 21
score on a scale | -2.21 (5.90) | -0.10 (7.49) | 0.14 (8.24)

11. Primary Outcome: Change in Survivor PTSD Symptom Severity at 3 Months Post-baseline (Self Report)
Description: Sum score on PTSD Checklist-5 (PCL-5), completed by survivor in reference to past month. Range: 0-80; higher scores indicate greater severity of PTSD symptoms.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 17 | 19 | 21
score on a scale | -12.12 (17.54) | -16.58 (13.32) | -16.25 (13.32)

12. Primary Outcome: Survivor Provisional PTSD Diagnostic Status at 3 Months Post-baseline (Self Report)
Description: Provisional PTSD diagnostic status based on PTSD Checklist-5 (PCL-5), completed by survivor in reference to past month. Survivors will be considered to have a provisional diagnosis if the following items are rated as 2 = "Moderately" or higher: one Criterion B item (questions 1-5), one Criterion C item (questions 6-7), two Criterion D items (questions 8-14), and two Criterion E items (questions 15-20).
Time Frame: 3 months
Population: Participants were excluded if they did not complete the scale at 3 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 17 | 19 | 21
Participants | 8 | 5 | 9

13. Primary Outcome: Change in Survivor Stress at 3 Months Post-baseline (Self Report)
Description: Sum score on the Stress subscale of the Depression and Anxiety Stress Scales (DASS-21), completed by survivor in reference to past week. Range: 0 to 21; higher scores indicate greater stress.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 20 | 21
score on a scale | -1.66 (5.39) | -2.42 (3.56) | -1.38 (3.58)

14. Primary Outcome: Change in Supporter Stress at 3 Months Post-baseline (Self Report)
Description: Sum score on the Stress subscale of the Depression and Anxiety Stress Scales (DASS-21), completed by supporter in reference to past week. Range: 0 to 21; higher scores indicate greater stress.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 20 | 18 | 20
score on a scale | -2.15 (3.30) | -1.22 (3.32) | -0.65 (3.07)

15. Primary Outcome: Change in Survivor Perceived Relationship Quality at 3 Months Post-baseline (Self Report)
Description: Sum score on the Relationship Assessment Scale, completed by survivor. Range: 7 to 35; higher scores indicate greater relationship quality.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 20 | 21
score on a scale | -0.39 (2.50) | -1.60 (4.45) | -1.76 (4.12)

16. Primary Outcome: Change in Supporter Perceived Relationship Quality at 3 Months Post-baseline (Self Report)
Description: Sum score on the Relationship Assessment Scale, completed by supporter. Range: 7 to 35; higher scores indicate greater relationship quality.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 20 | 18 | 20
score on a scale | 0.35 (3.94) | 0.39 (2.00) | -2.10 (4.33)

17. Secondary Outcome: Survivor Willingness to Participate in Criminal Justice Process at 1 Month Post-baseline (Self Report)
Description: Sum score score on measure created for this study, completed by survivor. Range: 0 to 10; higher scores indicate greater willingness.
Time Frame: 1 month
Population: Participants were excluded if they did not complete this scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 21 | 21
score on a scale | -0.21 (1.69) | 0.57 (1.99) | -0.19 (1.33)

18. Secondary Outcome: Survivor Participation in Criminal Justice Process at 1 Month Post-baseline (Self Report)
Description: Mean score on measure created for this study, completed by survivor. Range: 0 to 1; higher scores indicate greater participation.
Time Frame: 1 month
Population: Participants were excluded if they did not complete this scale.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 21 | 21 | 21
score on a scale | 0.64 (0.07) | 0.49 (0.07) | 0.52 (0.07)

19. Secondary Outcome: Change in Survivor Depression at 3 Months Post-baseline (Self Report)
Description: Sum score on the Depression subscale of the Depression and Anxiety Stress Scales (DASS-21), completed by survivor in reference to past week. Range: 0 to 21; higher scores indicate greater depression.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 20 | 21
score on a scale | -1.58 (6.15) | -3.00 (3.15) | -2.52 (4.57)

20. Secondary Outcome: Change in Supporter Depression at 3 Months Post-baseline (Self Report)
Description: Sum score on the Depression subscale of the Depression and Anxiety Stress Scales (DASS-21), completed by supporter in reference to past week. Range: 0 to 21; higher scores indicate greater depression.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 20 | 18 | 20
score on a scale | -0.80 (2.88) | -0.72 (2.02) | 0.44 (4.05)

21. Secondary Outcome: Change in Survivor Anxiety at 3 Months Post-baseline (Self Report)
Description: Sum score on the Anxiety subscale of the Depression and Anxiety Stress Scales (DASS-21), completed by survivor in reference to past week. Range: 0 to 21; higher scores indicate greater anxiety.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 20 | 21
score on a scale | -1.53 (4.50) | -1.50 (3.22) | -2.10 (5.40)

22. Secondary Outcome: Change in Supporter Anxiety at 3 Months Post-baseline (Self Report)
Description: Sum score on the Anxiety subscale of the Depression and Anxiety Stress Scales (DASS-21), completed by supporter in reference to past week. Range: 0 to 21; higher scores indicate greater anxiety.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 21 | 21 | 21
score on a scale | 0.33 (1.53) | 1.00 (2.51) | 0.33 (1.53)

23. Secondary Outcome: Change in Survivor Role Impairment at 3 Months Post-baseline (Self Report)
Description: Sum score on Work/School/Responsibility Impairment subscale of the Behavioral Activation for Depression Scale (BADS), completed by survivor in reference to past week. Range: 0 to 30; higher scores indicate more impairment.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 20 | 21
score on a scale | -2.95 (6.97) | -3.75 (5.82) | -4.00 (5.02)

24. Secondary Outcome: Change in Survivor Social Impairment at 3 Months Post-baseline (Self Report)
Description: Sum score on Social Impairment subscale of the Behavioral Activation for Depression Scale (BADS), completed by survivor in reference to past week. Range: 0 to 30; higher scores indicate more impairment.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 20 | 21
score on a scale | -3.21 (6.60) | -0.40 (7.71) | -1.57 (7.72)

25. Secondary Outcome: Change in Survivor Flourishing at 3 Months Post-baseline (Self Report)
Description: Sum score on Flourishing Index Measure, completed by survivor. Range: 0 to 120; higher scores indicate more flourishing.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 19 | 21
score on a scale | 0.21 (16.70) | 2.89 (12.43) | -2.90 (13.43)

26. Secondary Outcome: Change in Supporter Flourishing at 3 Months Post-baseline (Self Report)
Description: Sum score on Flourishing Index Measure, completed by supporter. Range: 0 to 120; higher scores indicate more flourishing.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 1.65 (10.39) | 5.22 (9.52) | -7.33 (17.39)

27. Secondary Outcome: Survivor Distress Associated With Supporter Negative Reactions at 1 Month Post-baseline (Self Report)
Description: Mean score on ratings of distress associated endorsed items on Negative Reactions subscale of the Social Reactions Questionnaire - Shortened, completed by survivor in reference to supporter's reactions to survivor in past month. Range: 0 to 3; higher scores indicate more distress.
Time Frame: 1 month
Population: Participants were excluded if they did not complete this scale.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 21 | 21 | 21
score on a scale | 1.28 (0.28) | 1.50 (0.24) | 1.37 (0.23)

28. Secondary Outcome: Supporter Positive Reactions to Disclosure at 1 Month Post-baseline (Informant Report)
Description: Sum score on Positive Reactions subscale of the Social Reactions Questionnaire - Shortened, completed by survivor in reference to supporter's reactions in past month. Range: 0 to 16; higher scores indicate more frequent positive reactions.
Time Frame: 1 month
Population: Only assessed among survivors reporting past-month disclosure to the supporter
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 15 | 19 | 16
score on a scale | 8.56 (1.02) | 9.53 (0.85) | 8.56 (1.02)

29. Secondary Outcome: Change in Survivor Typical Alcohol Consumption (Quantity) at 3 Months Post-baseline (Self Report)
Description: Number of typical drinks per week in past month reported by survivor on the Daily Drinking Questionnaire
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 20 | 20
drinks per week | 0.58 (5.96) | -1.80 (2.89) | -0.25 (9.30)

30. Secondary Outcome: Change in Survivor Typical Alcohol Consumption (Frequency) at 3 Months Post-baseline (Self Report)
Description: Number of typical drinking days per week in past month reported by survivor on the Daily Drinking Questionnaire. Range: 0 to 7.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 20 | 20
days per week | 0.32 (1.60) | -0.40 (0.99) | 0.25 (1.65)

31. Secondary Outcome: Change in Survivor Typical Alcohol Consumption (Hours) at 3 Months Post-baseline (Self Report)
Description: Number of typical drinking hours per week in past month reported by survivor on the Daily Drinking Questionnaire.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: hours per week
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 19 | 20
hours per week | 1.32 (7.45) | -0.79 (3.87) | -1.95 (8.51)

32. Secondary Outcome: Supporter Perceived Helping Ineffectiveness at 1 Month Post-baseline (Self Report)
Description: Sum score on the Confusion subscale of the Impact on Friends measure, completed by supporter in reference to the past month. Range: 6 to 30; higher scores indicate greater perceived ineffectiveness.
Time Frame: 1 month
Population: Participants were excluded if they did not complete this scale.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 21 | 21 | 21
score on a scale | 12.13 (0.91) | 12.78 (0.90) | 14.57 (0.91)

33. Secondary Outcome: Supporter Distress in Helping at 1 Month Post-baseline (Self Report)
Description: Sum score on the Emotional Distress subscale of the Impact on Friends measure, completed by supporter in reference to the past month. Range: 24 to 120; higher scores indicate greater distress.
Time Frame: 1 month
Population: Participants were excluded if they did not complete this scale.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 21 | 21 | 21
score on a scale | 53.59 (2.82) | 55.99 (2.80) | 61.57 (2.83)

34. Secondary Outcome: Supporter Accommodation of Survivor PTSD Symptoms at 1 Month Post-baseline (Self Report)
Description: Sum score on the Significant Others' Responses to Trauma Scale (SORTS), completed by supporter in reference to the past month. Range: 0 to 112; higher scores indicate greater accommodation.
Time Frame: 1 month
Population: Participants were excluded if they did not complete this scale.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 12.78 (2.96) | 8.64 (2.95) | 17.66 (2.01)

35. Secondary Outcome: Change in Survivor Cannabis Use Frequency at 3 Months Post-baseline (Self Report)
Description: Number of days of cannabis use in past 2 weeks, as reported by survivor. Range: 0 to 14.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 19 | 21
Days | -0.11 (1.79) | 0.63 (2.39) | -1.62 (2.91)

36. Secondary Outcome: Change in Survivor Prescription Opioid Misuse Frequency at 3 Months Post-baseline (Self Report)
Description: Number of days of prescription opioid use not as prescribed in past 2 weeks, as reported by survivor. Range: 0 to 14.
Time Frame: Baseline, 3 months
Population: Analyses could not be performed because no participants reported opioid use.
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 0 | 0 | 0

37. Secondary Outcome: Change in Survivor Non-prescription Opioid Use Frequency at 3 Months Post-baseline (Self Report)
Description: Number of days of non-prescription opioid use in past 2 weeks, as reported by survivor. Range: 0 to 14.
Time Frame: Baseline, 3 months
Population: Analyses could not be performed because no participants reported non-prescription opioid use.
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 0 | 0 | 0

38. Secondary Outcome: Change in Survivor Prescription Amphetamine Misuse Frequency at 3 Months Post-baseline (Self Report)
Description: Number of days of prescription amphetamine use not as prescribed in past 2 weeks, as reported by survivor. Range: 0 to 14.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 19 | 21
Days | 0.11 (0.46) | -0.05 (0.23) | 0.24 (1.09)

39. Secondary Outcome: Change in Survivor Methamphetamine Use Frequency at 3 Months Post-baseline (Self Report)
Description: Number of days of methamphetamine use in past 2 weeks, as reported by survivor. Range: 0 to 14.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 21 | 21
Days | 0.16 (0.69) | 0.29 (1.31) | -0.19 (0.87)

40. Secondary Outcome: Change in Survivor Cigarette Use Frequency at 3 Months Post-baseline (Self Report)
Description: Number of days of cigarette use in past 2 weeks, as reported by survivor. Range: 0 to 14.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 19 | 21
Days | -0.05 (0.23) | -0.16 (0.37) | -0.10 (0.44)

41. Secondary Outcome: Change in Survivor Cigarette Use Quantity at 3 Months Post-baseline (Self Report)
Description: Number of cigarettes smoked in a typical day in past 2 weeks, as reported by survivor.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: Cigarettes Per Day
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 19 | 20 | 21
Cigarettes Per Day | -0.01 (0.05) | -1.05 (3.36) | -0.62 (2.62)

42. Other Pre Specified Outcome: Survivor Disclosure Frequency to Supporter at 1 Month Post-baseline (Informant Report)
Description: Single item representing frequency of survivor's disclosures to supporter in past month, completed by supporter, adapted from the Early Intervention Clinic Disclosure Scale. Participants were instructed to enter a numerical value corresponding to number of disclosures. Higher scores indicate more frequent disclosure.
Time Frame: 1 month
Population: Participants were excluded if they did not complete this item.
Measure: Mean (Standard Error); unit: disclosures
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors)
Number analyzed (Participants) | 21 | 21 | 21
disclosures | 2.56 (0.21) | 2.70 (0.21) | 2.02 (0.20)

43. Other Pre Specified Outcome: Supporter Negative Reactions to Disclosure at 1 Month Post-baseline (Self Report)
Description: Sum score on Negative Reactions subscale of the Social Reactions Questionnaire - Shortened, completed by supporter in reference to supporter's reactions to survivor in past month. Range: 0 to 48; higher scores indicate more frequent negative reactions.
Time Frame: 1 month
Population: Only assessed among supporters reporting past-month receipt of disclosure from the survivor
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 18 | 19 | 11
score on a scale | 2.22 (3.12) | 1.79 (2.20) | 4.19 (3.62)

44. Other Pre Specified Outcome: Supporter Positive Reactions to Disclosure at 1 Month Post-baseline (Self Report)
Description: Sum score on Positive Reactions subscale of the Social Reactions Questionnaire - Shortened, completed by supporter in reference to supporter's reactions to survivor in past month. Range: 0 to 16; higher scores indicate more frequent positive reactions.
Time Frame: 1 month
Population: Only assessed among supporters reporting past-month receipt of disclosure from the survivor
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 18 | 19 | 11
score on a scale | 8.56 (0.63) | 8.74 (0.69) | 9.36 (0.99)

45. Other Pre Specified Outcome: Survivor Perceived Cultural Responsiveness of Intervention at 1 Month Post-baseline (Self Report)
Description: Sum score on survey created for this study, completed by survivor. Range: 4 to 16; higher scores indicate greater perceived cultural responsiveness of intervention.
Time Frame: 1 month
Population: Participants were excluded if they did not complete this scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors)
Number analyzed (Participants) | 19 | 21
score on a scale | 9.84 (1.74) | 10.19 (1.99)

46. Other Pre Specified Outcome: Supporter Perceived Cultural Responsiveness of Intervention at 1 Month Post-baseline (Self Report)
Description: as for outcome 45
Time Frame: 1 month
Population: Participants were excluded if they did not complete this scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters)
Number analyzed (Participants) | 20 | 20
score on a scale | 10.35 (1.84) | 10.45 (1.76)

47. Other Pre Specified Outcome: Survivor Perceived Impact of Intervention at 1 Month Post-baseline (Self-report)
Description: Sum score on survey created for this study, completed by survivor. Range: 4 to 20; higher scores indicate greater perceived impact of intervention.
Time Frame: 1 month
Population: Participants were excluded if they did not complete this scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors)
Number analyzed (Participants) | 18 | 21
score on a scale | 16.56 (2.50) | 15.71 (2.37)

48. Other Pre Specified Outcome: Supporter Perceived Impact of Intervention at 1 Month Post-baseline (Self-report)
Description: Sum score on survey created for this study, completed by supporter. Range: 4 to 20; higher scores indicate greater perceived impact of intervention.
Time Frame: 1 month
Population: Participants were excluded if they did not complete this scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters)
Number analyzed (Participants) | 20 | 20
score on a scale | 16.80 (2.53) | 16.60 (2.19)

49. Other Pre Specified Outcome: Change in Supporter Typical Alcohol Consumption (Quantity) at 3 Months Post-baseline (Self Report)
Description: Number of typical drinks per week in past month reported by supporter on the Daily Drinking Questionnaire. Range: 0 to 7.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: Drinks Per Week
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 20 | 18 | 19
Drinks Per Week | 0.25 (2.59) | -0.78 (1.48) | -1.87 (5.99)

50. Other Pre Specified Outcome: Change in Supporter Typical Alcohol Consumption (Frequency) at 3 Months Post-baseline (Self Report)
Description: Number of typical drinking days per week in past month reported by supporter on the Daily Drinking Questionnaire. Range: 0 to 7.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: Days Per Week
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 20 | 18 | 19
Days Per Week | 0.05 (0.83) | -0.22 (0.69) | -0.21 (1.32)

51. Other Pre Specified Outcome: Change in Supporter Typical Alcohol Consumption (Hours) at 3 Months Post-baseline (Self Report)
Description: Number of typical drinking hours per week in past month reported by supporter on the Daily Drinking Questionnaire.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: Hours Per Week
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 20 | 18 | 19
Hours Per Week | 2.30 (8.90) | -0.89 (2.03) | -1.26 (7.09)

52. Other Pre Specified Outcome: Change in Supporter Cannabis Use Frequency at 3 Months Post-baseline (Self Report)
Description: Number of days of cannabis use in past 2 weeks, as reported by supporter. Range: 0 to 14.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 20 | 18 | 20
Days | 0.45 (1.88) | -0.11 (0.32) | -0.85 (3.56)

53. Other Pre Specified Outcome: Change in Supporter Prescription Opioid Misuse Frequency at 3 Months Post-baseline (Self Report)
Description: Number of days of prescription opioid use not as prescribed in past 2 weeks, as reported by supporter. Range: 0 to 14.
Time Frame: Baseline, 3 months
Population: It was not possible to compute change scores because no participants reported prescription opioid use at any assessment
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 0 | 0 | 0

54. Other Pre Specified Outcome: Change in Supporter Non-prescription Opioid Use Frequency at 3 Months Post-baseline (Self Report)
Description: Number of days of non-prescription opioid use in past 2 weeks, as reported by supporter. Range: 0 to 14.
Time Frame: Baseline, 3 months
Population: It was not possible to compute change scores because no participants reported non-prescription opioid use at any assessment
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 0 | 0 | 0

55. Other Pre Specified Outcome: Change in Supporter Prescription Amphetamine Misuse Frequency at 3 Months Post-baseline (Self Report)
Description: Number of days of prescription amphetamine use not as prescribed in past 2 weeks, as reported by supporter. Range: 0 to 14.
Time Frame: Baseline, 3 months
Population: It was not possible to compute change scores because amphetamine use was very low base rate
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 0 | 0 | 0

56. Other Pre Specified Outcome: Change in Supporter Methamphetamine Use Frequency at 3 Months Post-baseline (Self Report)
Description: Number of days of methamphetamine use in past 2 weeks, as reported by supporter. Range: 0 to 14.
Time Frame: Baseline, 3 months
Population: It was not possible to compute change scores because no participants reported methamphetamine use at any assessment
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 0 | 0 | 0

57. Other Pre Specified Outcome: Change in Supporter Cigarette Use Frequency at 3 Months Post-baseline (Self Report)
Description: Number of days of cigarette use in past 2 weeks, as reported by supporter. Range: 0 to 14.
Time Frame: Baseline, 3 months
Population: Because this is a change score, participants were excluded listwise if they had missing data at one or both assessments. It was not possible to compute change scores for the Supporter-only condition because no participants reported cigarette use.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 20 | 0 | 20
Days | -0.10 (0.31) |  | -0.15 (2.37)

58. Other Pre Specified Outcome: Change in Supporter Cigarette Use Quantity at 3 Months Post-baseline (Self Report)
Description: Number of cigarettes smoked in a typical day in past 2 weeks, as reported by supporter.
Time Frame: Baseline, 3 months
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: Cigarettes Per Day
Arm/Group | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
Number analyzed (Participants) | 20 | 0 | 20
Cigarettes Per Day | -0.05 (0.22) |  | -0.18 (1.16)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 3 months
Arm/Group | Dyadic CARE (Survivors) | Supporter-Only CARE (Survivors) | Waitlist Control (Survivors) | Dyadic CARE (Supporters) | Supporter-Only CARE (Supporters) | Waitlist Control (Supporters)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/21 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/21 | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-04-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT05345405/Prot_SAP_ICF_000.pdf